CLINICAL TRIAL: NCT05182164
Title: Combination of Pembrolizumab and Cabozantinib in Patients With Advanced Sarcomas
Acronym: PEMBROCABOSARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ipsen (Industry); MSD France (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB2020-02
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Soft Tissue Sarcoma Adult; Advanced Soft-tissue Sarcoma; Ewing Sarcoma; Osteosarcoma; Undifferentiated Pleomorphic Sarcoma
Keywords: soft-tissue sarcoma; immune checkpoint inhibitor
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma; Histiocytoma, Malignant Fibrous; Sarcoma | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: 3 independent sigle-arm, multicenter, phase II trials, based on 2-stage Simon's optimal design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stratum 1: advanced undifferentiated pleomorphic sarcoma (Experimental): Patients with advanced undifferentiated pleomorphic sarcoma will be treated by the combination of pembrolizumab + cabozantinib
  Interventions: Drug: Association of pembrolizumab + cabozantinib
- Stratum 2: advanced osteosarcoma (Experimental): Patients with advanced osteosarcoma will be treated by the combination of pembrolizumab + cabozantinib
  Interventions: Drug: Association of pembrolizumab + cabozantinib
- Stratum 3: advanced Ewing sarcoma (Experimental): Patients with advanced Ewing sarcoma will be treated by the combination of pembrolizumab + cabozantinib
  Interventions: Drug: Association of pembrolizumab + cabozantinib

INTERVENTIONS:
Drug: Association of pembrolizumab + cabozantinib — A treatment cycle consists of 3 weeks. Pembrolizumab will be administered intraveinously on day 1 every 3 weeks (200 mg).
  Cabozantinib will be administered per os, once daily (40 mg), and given on a continuous basis.

SUMMARY:
Phase II trial with three independent strata to independently assess the effects of the association of pembrolizumab and cabozantinib in advanced sarcomas.

DETAILED DESCRIPTION:
3 independent, multicenter, prospective, signel-arm phase II trial, based on 2-stage Simon's optimal design, will be conducted in parallel to assess the efficacy of pembrolizumab + cabozantinib, in distinct populations of sarcomas:

* stratum 1: advanced undiffenrentiated pleomorphic sarcoma
* stratum 2: advanced osteosarcoma
* stratum 3: advanced ewing sarcoma

ELIGIBILITY:
Inclusion Criteria:

1. Histology: undifferentiated pleomorphic sarcoma (stratum 1), bone osteosarcoma (stratum 2), bone or extraskeletal or Ewing sarcoma (stratum 3),
2. Advanced non resectable / metastatic disease,
3. Recurrent disease or progression after standard therapy,
4. Documented progression according to RECIST criteria.
5. Have provided tissue of a tumor lesion from < 3 months old archival tissue sample obtained on locally advanced disease, or metastatis with no subsequent treatment since or from a newly obtained core or excisional biopsy,
6. No more of three previous lines of systemic therapy for advanced disease,
7. Age ≥ 18 years,
8. Eastern Cooperative Oncology Group ≤ 1,
9. Measurable disease according to RECIST v1.1 outside any previously irradiated field. At least one site of disease must be uni-dimensionally ≥ 10 mm,
10. Life expectancy > 3 months,
11. Participant must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement,
12. No symptomatic central nervous system disease,
13. No chronic use of glucocorticoids.
14. Adequate hematological, renal, metabolic and hepatic function,
15. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
16. At least three weeks since last chemotherapy, immunotherapy and two weeks for any other pharmacological treatment and/or radiotherapy,
17. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia of any grade, non-painful peripheral neuropathy grade ≤ 2 and endocrine-related grade ≤ 2 requiring treatment or hormone replacement) (according to NCI-CTCAE, version 5.0). For patients previously treated by radiotherapy, they must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis,
18. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication. Both women and men must agree to use 2 medically acceptable methods of contraception throughout the treatment period and for 6 months after discontinuation of treatment. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥ 1 year,
19. Voluntary signed and dated written informed consents prior to any specific study procedure,
20. Patients with a social security in compliance with the French Law.

Exclusion Criteria:

1. Previous treatment with Pembrolizumab or Cabozantinib,
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumabor any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways),
3. Evidence of progressive or symptomatic central nervous system or leptomeningeal metastases,
4. Men or women of childbearing potential who are not using an effective method of contraception; women who are pregnant or breast feeding, men or women who are planning to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment,
5. Participation to a study involving a medical or therapeutic intervention in the last 21 days,
6. Previous enrolment in the present study,
7. Patient unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons,
8. Patient unable to swallow,
9. Known hypersensitivity to any involved study drug or of its formulation components,
10. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy is not considered a form of systemic treatment and is allowed.
11. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment,
12. History of idiopathic pulmonary fibrosis, history of non-infectious pneumonitis that required steroids, current pneumonitis/interstitial lung disease, drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted,
13. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
14. Has a known history of HIV infection and/or of active TB (Bacillus Tuberculosis),
15. Treatment with anticoagulants such as anti-Vitamin K, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel),
16. Previous allogenic bone marrow transplant or solid organ transplantation,
17. Has an active infection requiring systemic treatment at study entry,
18. The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before treatment. Note: if initial QTcF is found to be > 500 ms, two additional ECGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard,
19. The subject requires chronic concomitant treatment of strong CYP3A4 inducers
20. The subject has experienced any of the following: Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment, Hemoptysis of ≥ 2.5 mL of red blood within 3 months before the first dose of study treatment, Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment, The subject has radiographic evidence of cavitating pulmonary lesion(s), The subject has tumor in contact with, invading or encasing any major blood vessels, or The subject has evidence of tumor invading the GI tract, or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
21. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions which are fully described in the study protocol: Cardiovascular disorders, Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation, Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy,
22. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
23. Has an history or current evidence of any condition, therapy, or laboratory abnormality that might counfound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
24. The subject is planning to have oral surgery/invasive dental procedure within the projected duration of the study, starting with the screening visit through 3 months after the last dose of study treatment or had such a procedure within 3 months of first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy of pembrolizumab and cabozantinib (independently for each stratum) | 6 months
  Efficacy will be assessed in terms of non-progression rate at 6 months and is defined as the proportion of patients with complete response (CR), or partial response (PR), or stable disease (SD) at 6 months from the start of the treatment, based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Best overall response, independently for each stratum | Throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best response across all time points (RECIST 1.1). The best overall response is determined once all the data for the patient is known (RECIST 1.1).
1-year progression-free survival, independently for each stratum | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first.
1-year overall survival, independently for each stratum | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
Safety profile, independently for each stratum: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5.
6-months non-progression rate according to iRECIST | 6 months
  Efficacy will be assessed in terms of non-progression rate at 6 months and is defined as the proportion of patients with complete response (CR), or partial response (PR), or stable disease (SD) at 6 months from the start of the treatment, based on iRECIST criteria (Seymour, 2017).
Blood cytokines levels | baseline, cycle 2 day 1, cycle 2 day 8, cycle 3 day 1, cycle 4 day 1, cycle 6 day 1 and at progression (each cycle is 21 days)
  Levels of cytokines in blood will be measured by ELISA.
Blood lymphocytes levels | baseline, cycle 2 day 1, cycle 2 day 8, cycle 3 day 1, cycle 4 day 1, cycle 6 day 1 and at progression (each cycle is 21 days)
  Levels of lymphocytes in blood will be measured by flow cytometry.
Blood kynurenine levels | baseline, cycle 2 day 1, cycle 2 day 8, cycle 3 day 1, cycle 4 day 1, cycle 6 day 1 and at progression (each cycle is 21 days)
  Levels of kynurenine in blood will be measured by ELISA.
Tumor immune cells levels | before treatment onset and cycle 2 day 8 (each cycle is 21 days)
  Levels of immune cells in tumor will be measured by immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital La Timone, Marseille
  - Institut Curie, Paris
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - IUCT Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif